CLINICAL TRIAL: NCT03604237
Title: Concordance Rate of Pathology Between Targeted Forceps Biopsy and Resected Specimen for Large Colorectal Tumors
Brief Title: Targeted Forceps Biopsy for Colorectal Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Eun Soo Kim, MD, PhD, Professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: KNUH201804
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Colorectal Neoplasms
Keywords: forceps biopsy; colorectal tumors
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeted forceps biopsy (Experimental): In this group, an endoscopist takes a forceps biopsy at depressed mucosa or large nodular area of large colorectal tumors after meticulous surface evaluation.
  Interventions: Diagnostic Test: Targeted group
- Conventional forceps biopsy (No Intervention): In this group, an endoscopist takes a forceps biopsy at the most convenient area of large colorectal tumors.

INTERVENTIONS:
Diagnostic Test: Targeted group — Forceps biopsy is taken after surface evaluation of the large colorectal tumors.
  Arms: Targeted forceps biopsy

SUMMARY:
This study evaluates whether targeted forceps biopsy with careful tumor surface evaluation can improve diagnostic accuracy of colorectal tumors larger than 2 cm during colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with colorectal neoplasms of the size larger than 2 cm

Exclusion Criteria:

* Patients who deny the participation in the study

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-08-01 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
pathologic diagnosis | 7 days
  The pathologic diagnosis of forceps biopsy is compared with the pathologic diagnosis of resected specimen of the colorectal tumor.

CONTACTS AND LOCATIONS:
Locations (1):
- Kyungpook National University Hospital, Daegu, South Korea